CLINICAL TRIAL: NCT06406673
Title: A Phase II Clinical Study of Cadonilimab(PD-1/CTLA-4 Bi-Specific Antibody) in Treatment-naïve or Relapsed Extensive Small Cell Lung Cancer
Brief Title: A Phase II Clinical Study of Cadonilimab in Treatment-naïve or Relapsed Extensive Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-SCLC-01
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-09

CONDITIONS: Extensive Small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort_1 (Experimental): Cohort_1 patients with no history of previous systemic treatment for ES-SCLC received cadonilimab with EC/EP and received concurrent palliative RT.
  Interventions: Drug: Cadonilimab+EC/ET+RT
- Cohort_2 (Experimental): Cohort_2 patients with recurrent SCLC and after at most one systemic treatment received cadonilimab plus vorolanib.
  Interventions: Drug: Cadonilimab+vorolanib

INTERVENTIONS:
Drug: Cadonilimab+EC/ET+RT — Cohort_1 patients with no history of previous systemic treatment for ES-SCLC received cadonilimab with EC/EP for two cycles (induction phase), then, those who did not progress received concurrent palliative RT and two cycles of cadonilimab with EC/EP (combination phase). Afterward they received cadonilimab every 3 weeks for a maximum of 2 years after study enrolment (maintenance phase).
  Arms: Cohort_1
Drug: Cadonilimab+vorolanib — Cohort_2 patients with recurrent SCLC and after at most one systemic treatment received cadonilimab plus vorolanib, until disease progression or unacceptable toxicity.
  Arms: Cohort_2

SUMMARY:
Small cell lung cancer (SCLC) accounts for 15% of lung cancer cases and is an aggressive cancer characterized by rapid growth, early metastasis, and a poor prognosis. Approximately 75% of SCLC patients present with extensive-stage disease at the time of diagnosis, which is classically defined as a disease that cannot be encompassed by a single radiation field. Before the era of immunotherapy, the standard first-line therapy for ES-SCLC was platinum-based chemotherapy with etoposide; Once complete remission (CR) or partial remission (PR) was achieved after chemotherapy, consolidative thoracic radiation was recommended. Despite this standard treatment, the median overall survival (OS) of ES-SCLC is about 8-11 months, which has not changed for about 40 years. Combining concurrent radiotherapy of the thorax and immunochemotherapy may have a synergistic effect.

Besides, for patients with recurrent SCLC, topotecan remains the only approved second-line treatment, and the outcomes are poor. With the most recent approval of EP plus a programmed death ligand 1(PD-L1) inhibitor, there are now more therapeutic options for managing ES-SCLC.The best second-line therapy after combination of chemo-immunotherapy is not well defined, as many second-line therapies were studied only after use of EP. However, second-line treatment options for patients with relapsed ES-SCLC are limited and include reintroduction of EP (with or without an immunotherapy), lurbinectedin, and topotecan.

Therefore, we designed this trial to explore the efficacy and safety of cadonilimab as second-line therapy for ES-SCLC. We present a safety profile and a final analysis of ORR.

In this single-center phase 2 trial, Cohort_1 patients with no history of previous systemic treatment for ES-SCLC received cadonilimab with EC/EP for two cycles (induction phase), then, those who did not progress received concurrent palliative RT and two cycles of cadonilimab with EC/EP (combination phase). Afterward they received cadonilimab every 3 weeks for a maximum of 2 years after study enrolment (maintenance phase). Cohort_2 patients with recurrent SCLC and after at most one systemic treatment received cadonilimab plus vorolanib, until disease progression or unacceptable toxicity.

The primary endpoints was objective response rate (ORR); the second endpoints were progression-free survival (PFS), disease control rate (DCR), overall survival (OS) and treatment-emergent adverse event (TEAE) .

ELIGIBILITY:
Inclusion Criteria:

1. All subjects voluntarily participated in the study and signed informed consent;
2. Male or female aged ≥18 years ;
3. Expected survival time ≥3 months;
4. ECOG 0-1;
5. Patients with extensive-stage small-cell Lung cancer confirmed by histopathology and/or cytology (according to Veterans Administration Lung Study Group (VALG) staging); 5-1）Cohort_1 patients who have not received any previous systemic anti-tumor therapy for extensive-stage small cell lung cancer, and included all patients with ≤5 extrapulmonary metastases.

   5-2）Cohort_2 patients with previous failure or intolerance to standard therapy for extensive-stage small cell lung cancer and received at most one systemic treatment:

   a) Those who have previously failed first-line platinum-based chemotherapy combined with immune checkpoint inhibitors, and have received at most one systemic treatment, as follows:
   * Receiving less than 2 lines of systemic therapy in the advanced stage of the disease;

     ②Immune checkpoint inhibitors include atezolizumab, durvalumab, slulimumab, adebelimab, etc.;

     ③Disease progression confirmed by imaging during or after the latest treatment b) Those who have only received first-line platinum-containing drug treatment in the past and failed, and have not received immune checkpoint inhibitor treatment, as follows:
   * Receiving less than 2 lines of systemic therapy in the advanced stage of the disease; ② The first-line treatment must be platinum-containing chemotherapy; ③ Disease progression confirmed by imaging during or after the latest treatment
6. Consent to provide archival tumor tissue specimens (10 unstained sections (anti-slip) surgical specimens (thickness 4-5μm)) or fresh tissue samples from primary or metastatic lesions within 3 years. If participants cannot provide tumor tissue samples, they can be enrolled if they meet other inclusion and exclusion criteria, after the evaluation of the investigator;
7. Must have at least one measurable lesion according to RECIST v1.1 definition; Lesions that had been previously treated with radiation could be included in a measurable lesion only if there was definite disease progression after radiation therapy.
8. Organ function level must meet the following criteria： 8-1) Blood routine: hemoglobin (HGB) ≥ 90g/L; Absolute neutrophil count (NEUT) ≥ 1.5×10 9 /L; Platelet count (PLT) ≥ 100×10 9 /L; 8-2) Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula).

   8-3) Liver function: total bilirubin (TBIL≤1.5 ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were all ≤2.5 ULN, and AST and ALT were both ≤5.0 ULN when liver metastasis was present; 8-4) coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5ULN; 8-5) no severe cardiac dysfunction with left ventricular ejection fraction ≥50%; 8-6) proteinuria ≤2+ or ≤1000mg/24h; 8-7) Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic laboratory abnormalities such as ALP elevation, hyperuricemia, and hyperglycemia, as judged by the investigator, and toxicity without safety risk, such as alopecia, grade 2 peripheral neurotoxicity, or decreased hemoglobin ≥90g/L, as judged by the investigator); 8-8) For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the start of treatment, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the whole treatment cycle and for 6 months after the end of treatment.
9. Women of reproductive age should agree to use effective contraception during the study period and for six months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating; Men should agree to use contraception during the study period and for six months after the study period ends;
10. Patients will be able to communicate well with the investigator, understand and comply with the requirements of the study.

Exclusion Criteria:

1. Histologically or cytologically confirmed NSCLC;
2. Previous medications:For Cohort_1: Exclude those who have received systemic anti-tumor therapy or with >5 extrapulmonary metastases; For Cohort_2: Those who have received more than one systemic treatment regimen
3. Participated in other domestic unapproved or unmarketed drug clinical trials and accepted the corresponding experimental drug treatment within 4 weeks before enrollment;
4. Imaging during the screening period shows that the tumor surrounds important blood vessels or has obvious necrosis or cavities, and the researcher determines that entering the study will cause a risk of bleeding(Only for Cohort_2).
5. Received any surgery or invasive treatment or operation within 4 weeks before enrollment (excluding intravenous catheterization, puncture drainage, puncture biopsy, etc.)
6. The patient currently has central nervous system (CNS) metastases or active brain or meningeal metastases. Treated subjects with BMS were required to meet the following criteria: asymptomatic; No radiographically demonstrated progression ≥4 weeks after completion of treatment; Completion of treatment ≥14 days before the first dose of the study drug; Systemic corticosteroid therapy (> 10mg/ day prednisone or equivalent) is not required for ≤14 days prior to the first dose of the study drug
7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
8. Any other medical condition, clinically significant metabolic abnormality, physical abnormality, or laboratory abnormality that, in the investigator's judgment, reasonably suspects the patient to have a medical condition or condition that is not suitable for the use of the study drug (such as having seizures that require treatment), or that would affect the interpretation of the study results, or put the patient at high risk;
9. Have received or plan to receive live attenuated vaccine within 4 weeks prior to initial administration;
10. Currently receiving anti-HBV treatment;
11. Received approved or under development systematic anti-tumor therapy within 28 days before enrollment;
12. Those who are known to be allergic to the active ingredient or excipients of the drug in this study;
13. Women who are pregnant (positive pregnancy test before medication) or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Overall survival (OS) | 24 months
  The OS is defined as the time from study entry to death from any cause.
Treatment-Emergent Adverse Event (TEAE) | 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No